CLINICAL TRIAL: NCT04725201
Title: Prospective Study on the Role of Intravenous Unfractionated Heparin Following Digital Replantation and Revascularization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-9178
Record Dates: First submitted 2021-01-09; First posted 2021-01-26 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Amputation; Traumatic, Hand
Keywords: Replantation; Revascularization; Unfractionated heparin; Finger
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Prospective randomized double-blinded clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous unfractionated heparin (Experimental): Administration of intravenous unfractionated heparin according to the Centre hospitalier de l'Université de Montréal (CHUM) deep vein thrombosis (DVT) protocol for 5 days after vascular anastomosis. A bolus will be administered intraoperatively based on the patient's weight. Dosages will be adjusted according to the activated partial thromboplastin time (aim for an APTT of 50-70), which will be measured 6 hours after the start of the protocol and after every dosage adjustment or every morning at 6 a.m. if no adjustments were made in the last 6 hours.
  Interventions: Drug: Intravenous unfractionated heparin
- Control (Sham Comparator): No administration of intravenous unfractionated heparin. These patients receive 5000 IU BID of heparin subcutaneously, as a standard post-operative protocol for all in-patients.
  The control group receives sham bolus intraoperatively of normal saline and a post-operative normal saline infusion at a fixed dose through an infusion pump to mimic IV heparin infusion.
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: Intravenous unfractionated heparin — See experimental arm description for intervention description.
  Arms: Intravenous unfractionated heparin
Drug: Sham — See sham comparator arm description for intervention description.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effectiveness of therapeutic dose intravenous heparin at improving replantation/revascularization success and its indications (if any) in participants who have suffered traumatic digital amputation. Digital replantation/revascularization success will be assessed in participants who receive continuous intravenous drip of thromboprophylactic heparin at a therapeutic dose (i.e. modifies INR to the desired range) contrasted to those who do not receive therapeutic dose heparin (i.e. does not modify INR to the desired range). In the study, replantation/revascularization success is defined as a clearly viable digit at the time of discharge. Secondary objectives include assessing postoperative complications associated with heparin use, such as bleeding, hematoma or heparin induced thrombocytopenia. The investigators would also assess the impact of categorical variables such as smoking status, mechanism of injury and comorbidities, on digital survival.

ELIGIBILITY:
Inclusion Criteria:

* All replantation and revascularization patients who are accepted into the CEVARMU program at the Centre hospitalier de l'Université de Montréal

Exclusion Criteria:

* Patients on anticoagulants, other than ASA, prior to admission (i.e. Coumadin, Eliquis, Pradaxa, Plavix, or similar medications)
* Patients with a contraindication for heparin (e.g. coagulopathy, acute ulcers, thrombocytopenia, severe liver damage, shock)
* Patients who suffered an amputation in the level of the carpal tunnel and proximal to it
* Patients who experienced a degloving injury

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2024-09-24 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Success of digit replantation or revascularization | Up to 14 days
  Success is defined as a clearly viable digit, determined by saturation with a pulse oximeter or by bleeding on needle pinprick.

SECONDARY OUTCOMES:
Heparin-related complications | Up to 14 days
  Complications include but are not limited to bleeding at or away from site of injury, hematoma, heparin-induced thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Mastropasqua, MD FRCSC, Principal Investigator — Université de Montréal
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No